CLINICAL TRIAL: NCT03812510
Title: A Phase 3 Open Label Safety Study of A-101 Topical Solution for the Treatment of Common Warts
Brief Title: Safety Study of A-101 Topical Solution for the Treatment of Common Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-101-WART-303
Record Dates: First submitted 2019-01-10; First posted 2019-01-23 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Common Wart
Keywords: common warts
MeSH Terms: conditions — Warts | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- A-101 (Experimental): Topical Solution
  Interventions: Drug: A-101

INTERVENTIONS:
Drug: A-101 — hydrogen peroxide topical solution 45%
  Other Names: hydrogen peroxide 45%

SUMMARY:
A Phase 3 Study of A-101 Topical Solution Applied Twice a Week in Subjects with Common Warts

DETAILED DESCRIPTION:
A Phase 3 Open Label Safety Study of A-101 Topical Solution for the Treatment of Common Warts

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal guardian is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
* Subject must have completed study participation in either A-101-WART-301 or A-101-WART-302.
* Male or female ≥ 1 years old.
* Subject has a clinical diagnosis of common warts (verruca vulgaris).
* Identified warts must have a longest axis of ≤8 mm

Exclusion Criteria:

* Subject has clinically atypical warts.
* Subject is immunocompromised
* Subject has a history of Human Immunodeficiency Virus (HIV) infection.
* Subject has had any Human Papilloma Virus (HPV) vaccine within 6 months prior to Visit 1.
* Subject has used any of the following intralesional therapies within the specified period prior to Visit 1:

  1. Immunotherapy (e.g., Candida antigen, mumps antigen, Trichophyton antigen); 8 weeks
  2. Anti-metabolite therapy (e.g., bleomycin, 5-fluorouracil); 8 weeks
* Subject has used any of the following systemic therapies within the specified period prior to Visit 1:

  1. Immunomodulatory/immunosuppressant therapy (e.g., etanercept, alefacept, infliximab); 16 weeks
  2. Glucocorticosteroids (inhaled and intra-nasal steroids are permitted); 28 days
* Subject has used any of the following topical therapies within the specified period prior to Visit 1 on or in the proximity to any of the common warts identified for treatment that in the investigator's opinion interferes with the study medication treatment or the study assessments:

  1. LASER, light or other energy-based therapy (e.g., intense pulsed light [IPL], photodynamic therapy [PDT]); 180 days
  2. Immunotherapy (e.g., imiquimod, squaric acid dibutyl ester [SADBE], etc.) 12 weeks
  3. Liquid nitrogen, electrodesiccation, curettage; 60 days
  4. Hydrogen peroxide; 90 days (other than IP from the 301/302 study)
  5. Antimetabolite therapy (e.g., 5-fluorouracil); 8 weeks
  6. Retinoids; 90 days
  7. Over-the-counter (OTC) wart therapies and cantharidin; 28 days
* Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in a proximity to any of the common warts identified for treatment that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

  1. Cutaneous malignancy; 180 days
  2. Sunburn; currently
  3. Pre-malignancy (e.g., actinic keratosis); currently
* Subject has a history of sensitivity to any of the ingredients in the study medications.
* Subject has any current skin or systemic disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations.
* Participation in another therapeutic investigational drug/device trial (other than the Aclaris 301 or 302 study) in which administration of an investigational treatment occurred within 30 days prior to Visit 1.
* Subject has an active malignancy.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gordon, MB, ChB, Study Director — Aclaris Therapeutics
Locations (43):
- United States (43):
  - Aclaris Investigational Site, Mobile, Alabama
  - Aclaris Investigational Site, Glendale, Arizona
  - Aclaris Investigational Site, Fort Smith, Arkansas
  - Aclaris Investigational Site, Hot Springs, Arkansas
  - Aclaris Investigational Site, Encinitas, California
  - Aclaris Investigational Site, Fountain Valley, California
  - Aclaris Investigational Site, San Diego, California
  - Aclaris Investigational Site, Denver, Colorado
  - Aclaris Investigational Site, Aventura, Florida
  - Aclaris Investigational Site, Jacksonville, Florida
  - Aclaris Investigational Site, Miami, Florida
  - Aclaris Investigational Site, Ocala, Florida
  - Aclaris Investigational Site, Newnan, Georgia
  - Aclaris Investigational Site, Indianapolis, Indiana
  - Aclaris Investigational Site, New Albany, Indiana
  - Aclaris Investigational Site, Louisville, Kentucky
  - Aclaris Investigational Site, Rockville, Maryland
  - Aclaris Investigational Site, Fridley, Minnesota
  - Aclaris Investigational Site, Saint Joseph, Missouri
  - Aclaris Investigational Sites, Omaha, Nebraska
  - Aclaris Investigational Site, Las Vegas, Nevada
  - Aclaris Investigational Site, Verona, New Jersey
  - Aclaris Investigational Site, Rochester, New York
  - Aclaris Investigational Site, Raleigh, North Carolina
  - Aclaris Investigational Site, Beachwood, Ohio
  - Aclaris Investigational Site, Bexley, Ohio
  - Aclaris Invesgational Site, Broomall, Pennsylvania
  - Aclaris Investigational Site, Fort Washington, Pennsylvania
  - Aclaris Investigational Site, Upper Saint Clair, Pennsylvania
  - Aclaris Investigational Site, Anderson, South Carolina
  - Aclaris Investigational Site, Charleston, South Carolina
  - Aclaris Investigational Site, Fountain Inn, South Carolina
  - Aclaris Investigational Site, Knoxville, Tennessee
  - Aclaris Investigational Site, Nashville, Tennessee
  - Aclaris Investigational Site, Arlington, Texas
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigational Site, College Station, Texas
  - Aclaris Investigational Site, Houston, Texas
  - Aclaris Investigational Site, Pflugerville, Texas
  - Aclaris Investigational Site, San Antonio, Texas
  - Aclaris Investigational Site, Lynchburg, Virginia
  - Aclaris Investigational Site, Norfolk, Virginia
  - Aclaris Investigational Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies.
Pre-assignment Details: In the A-101-WART-303 study, subjects will be followed every 6 weeks to assess for a recurrence or development of new common warts. If a recurrence occurs or a new wart develops these subjects may return to the site to receive A-101 Topical Solution 45% twice a week for an additional treatment cycle of 8 weeks.
Period: Overall Study
Arm/Group | A-101
Started | 426
Completed | 274
Not Completed | 152
Not completed — Lost to Follow-up | 39
Not completed — Withdrawal by Subject | 42
Not completed — Physician Decision | 2
Not completed — Study Terminated by Sponsor | 9
Not completed — Did Not Start Study Medication | 55
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Groups:
- A-101 Hydrogen Peroxide Topical Solution 45%: In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies. However, Baseline Measures were collected as a single arm for the study.
Arm/Group | A-101 Hydrogen Peroxide Topical Solution 45%
Number analyzed (Participants) | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (18.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253
  Male | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55
  Not Hispanic or Latino | 346
  Unknown or Not Reported | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 396
  More than one race | 0
  Unknown or Not Reported | 7
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 18
  II - Burns Easily | 132
  III - Burns Moderately | 177
  IV - Burns Minimally | 75
  V - Rarely Burns | 16
  VI - Never Burns | 8
Total Warts Treated [Count of Participants; unit: Participants]
  0 | 56
  1 | 214
  2 | 65
  3 | 24
  4 | 27
  5 | 15
  6 | 25
Does the Subject have a Common Wart at Entry to Open-Label Study? [Count of Participants; unit: Participants]
  Yes | 370
  No | 56
Longest Axis of Largest Wart Treated [Mean (Standard Deviation); unit: millimetres] — Population: 56 subjects did not have a Wart when they entered the open label extension study.
  millimetres
    number analyzed (Participants) | 370
    (all) | 4.5 (1.63)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Treatment Emergent AEs After Application of A-101 45% for the Treatment of Common Warts
Description: Safety exposure will be measured by the proportion of subjects exposed to A-101 45% who have emergent adverse events. In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies. In the A-101-WART-303 study, subjects will be followed every 6 weeks to assess for a recurrence or development of new common warts. If a recurrence occurs or a new wart develops these subjects may return to the site to receive A-101 Topical Solution 45% twice a week for an additional treatment cycle of 8 weeks.
Time Frame: Baseline to a maximum of 341 days
Population: The amount of patients in the various treatment cycles differs because patients without wart recurrences or new warts developing may not return for additional treatment cycles.
Measure: Count of Participants; unit: Participants
Groups:
- A-101 45% (Active): Topical solution, hydrogen peroxide 45% A-101: hydrogen peroxide 45% topical solution
- Isopropyl Alcohol and Water (Vehicle): Topical solution, isopropyl alcohol and water Vehicle: Vehicle solution containing isopropyl alcohol and water
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 163 | 213
Participants | 70 | 116

2. Secondary Outcome: Durability of Response: Median Number of Days All Warts Remain Clear by Treatment Group and Treatment Cycle for Subjects With All Warts Achieving a Status of Clear (PWA=0) (Treatment Cycle 1)
Description: Safety exposure will be measured by the proportion of subjects exposed to A-101 45% who have emergent adverse events. In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies.
  This endpoint measures the durability of response by time to wart recurrence by prior study treatment group in the Safety Population.
Time Frame: Baseline to a maximum of 207 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 163 | 213
days | 207 [132 to 207] | 153 [149 to 153]

3. Secondary Outcome: Durability of Response: Median Number of Days All Warts Remain Clear by Treatment Group and Treatment Cycle for Subjects With All Warts Achieving a Status of Clear (PWA=0) (Treatment Cycle 2)
Description: Safety exposure will be measured by the proportion of subjects exposed to A-101 45% who have emergent adverse events. In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies.
  Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Baseline to a maximum of 248 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 118 | 139
days | NA [NA to NA] — A median, and upper and lower limits of the Confidence Interval were not able to be calculated in the Active group due to an insufficient number of participants with events. | NA [67 to NA] — A median and upper limit of the Confidence Interval were not able to be calculated in the Vehicle group due to an insufficient number of participants with events.

4. Secondary Outcome: Durability of Response: Median Number of Days All Warts Remain Clear by Treatment Group and Treatment Cycle for Subjects With All Warts Achieving a Status of Clear (PWA=0) (Treatment Cycle 3)
Description: as for outcome 3
Time Frame: Baseline to a maximum of 290 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 34 | 30
days | NA [22 to NA] — A median and upper limit of the Confidence Interval were not able to be calculated in the Active group due to an insufficient number of participants with events. | NA [NA to NA] — A median, and lower and upper limits of the Confidence Intervals were not able to be calculated in the Vehicle group due to an insufficient number of participants with events.

5. Secondary Outcome: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale (Treatment Cycle 1)
Description: as for outcome 3
Time Frame: Baseline to a maximum of 207 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 147 | 177
percentage of wart clearance | 19.90 (36.590) | 24.92 (34.489)

6. Secondary Outcome: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale (Treatment Cycle 2)
Description: as for outcome 3
Time Frame: Baseline to a maximum of 248 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 107 | 114
percentage of wart clearance | 24.92 (39.240) | 22.37 (39.513)

7. Secondary Outcome: Mean Per-Subject Percent of All Warts That Were Clear on the Physician Wart Assessment (PWA) Scale (Treatment Cycle 3)
Description: as for outcome 3
Time Frame: Baseline to a maximum of 290 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 31 | 29
percentage of wart clearance | 30.91 (43.205) | 15.52 (32.407)

8. Secondary Outcome: Mean Per-Subject Percent Wart Clearance for Subjects With Single Wart at Baseline by Treatment Group and Treatment Cycle (Treatment Cycle 1)
Description: Safety exposure will be measured by the proportion of subjects exposed to A-101 45% who have emergent adverse events. In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies.
  Median time to achieve onset of Clearance (PWA=0) for all treated warts. Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Baseline to a maximum of 207 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 87 | 107
percent of wart clearance | 13 (14.94) | 13 (12.15)

9. Secondary Outcome: Mean Per-Subject Percent Wart Clearance for Subjects With Single Wart at Baseline by Treatment Group and Treatment Cycle (Treatment Cycle 2)
Description: as for outcome 8
Time Frame: Baseline to a maximum of 248 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 62 | 66
percent of wart clearance | 12 (19.35) | 13 (19.70)

10. Secondary Outcome: Mean Per-Subject Percent Wart Clearance for Subjects With Single Wart at Baseline by Treatment Group and Treatment Cycle (Treatment Cycle 3)
Description: as for outcome 8
Time Frame: Baseline to a maximum of 290 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of wart clearance
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 23 | 20
percent of wart clearance | 7 (30.43) | 1 (5.00)

11. Secondary Outcome: Time to Clearance of All Warts Warts by Treatment Group and Treatment Cycle (Treatment Cycle 1)
Description: Safety exposure will be measured by the proportion of subjects exposed to A-101 45% who have emergent adverse events. In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies.
  The median was unable to be calculated, so the 25th percentile was used as the time to achieve onset of Clearance (PWA=0) for all treated warts. Efficacy will be assessed using the Physician's Wart Assessment Scale (PWA) which is a 4 point scale. A higher amount of warts cleared represents a better outcome.
Time Frame: Baseline to a maximum of 207 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 163 | 213
days | 70 [66 to 182] | NA [64 to NA] — The upper limit of the Confidence Interval was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.

12. Secondary Outcome: Time to Clearance of All Warts Warts by Treatment Group and Treatment Cycle (Treatment Cycle 2)
Description: as for outcome 8
Time Frame: Baseline to a maximum of 248 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 118 | 137
days | 156 [137 to NA] — The upper limit of the 95% Confidence Interval was not able to be calculated in the Active group due to an insufficient number of participants with events. | NA [147 to NA] — The upper limit of the 95% Confidence Interval was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.

13. Secondary Outcome: Time to Clearance of All Warts Warts by Treatment Group and Treatment Cycle (Treatment Cycle 3)
Description: as for outcome 8
Time Frame: Baseline to a maximum of 290 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | A-101 45% (Active) | Isopropyl Alcohol and Water (Vehicle)
Number analyzed (Participants) | 34 | 30
days | NA [78 to NA] — A median and upper limit of the Confidence Interval were not able to be calculated in the Active group due to an insufficient number of participants with events. | 124 [124 to NA] — An upper limit of the Confidence Interval was not able to be calculated in the Vehicle group due to an insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: 182 days. The investigator must start reporting non-serious AEs starting with the subject's first study medication treatment continuing until the subject's last study visit.
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and that did not necessarily have a causal relationship with the study medication.
  Safety summaries by study medication group will include listings by study medication of adverse events incidences within each MedDRA System Organ Class, and changes from pre-application values in vital signs.
Groups:
- A-101 A-101: Hydrogen Peroxide Topical Solution 45%: In order to be eligible for A-101-WART-303, subjects must have completed protocol treatment on either the A-101-WART-301 or A-101-WART-302 study. The A-101-WART-303 study was an open-label with a single arm where all subjects received A-101 Topical Solution 45% twice a week. Since A-101-WART-303 is an extension study, statistical analyses were performed by stratifying patients by treatment arms in the A-101-WART-301 or A-101-WART-302 studies. However, Baseline Measures were collected as a single arm for the study.
Arm/Group | A-101 A-101: Hydrogen Peroxide Topical Solution 45%
All-Cause Mortality (participants affected / at risk) | 0/376
Serious Adverse Events (participants affected / at risk) | 1/376
Other Adverse Events (participants affected / at risk) | 186/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 A-101: Hydrogen Peroxide Topical Solution 45% (N=376)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 A-101: Hydrogen Peroxide Topical Solution 45% (N=376)
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Goitre (Endocrine disorders) | 1 (1)
Meibomian gland dysfunction (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Application site dermatitis (General disorders) | 1 (1)
Application site discomfort (General disorders) | 1 (1)
Application site dryness (General disorders) | 1 (1)
Application site erosion (General disorders) | 5 (5)
Application site erythema (General disorders) | 13 (13)
Application site irritation (General disorders) | 1 (1)
Application site laceration (General disorders) | 1 (1)
Application site oedema (General disorders) | 1 (1)
Application site pain (General disorders) | 131 (131)
Application site pallor (General disorders) | 20 (20)
Application site papules (General disorders) | 1 (1)
Application site paraesthesia (General disorders) | 1 (1)
Application site pruritus (General disorders) | 40 (40)
Application site scab (General disorders) | 19 (19)
Application site swelling (General disorders) | 1 (1)
Application site vesicles (General disorders) | 4 (4)
Peripheral swelling (General disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Application site infection (Infections and infestations) | 27 (27)
Bronchitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 2 (2)
Gastroenteritis (General disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3)
Hordeolum (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Otitis externa (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Urinary tract infection (General disorders) | 2 (2)
Viral upper respiratory tract infection (General disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (General disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (General disorders) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Back pain (Metabolism and nutrition disorders) | 3 (3)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 7 (7)
Sciatica (Nervous system disorders) | 1 (1)
Embedded device (Product Issues) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4 (4)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT03812510/Prot_000.pdf
  • Informed Consent Form (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03812510/ICF_001.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03812510/SAP_002.pdf